CLINICAL TRIAL: NCT05438199
Title: Prototyping a Device for Automating Stool and Urine Output Tracking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00104899
Record Dates: First submitted 2022-06-17; First posted 2022-06-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Waste Output
Keywords: urine output; stool output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- apparatus use (Experimental): All participants will use the apparatus following the same procedures. They will weigh themselves on a scale located in the bathroom, use the apparatus with or without "hats" ("hats" refer to a plastic container used to catch stool/urine that needs to be placed between the toilet rim and the toilet seat and discarded after each use) and weigh themselves after using the toilet.
  Interventions: Device: Toilet seat that measures waste output

INTERVENTIONS:
Device: Toilet seat that measures waste output — Participants will use a toilet that includes a apparatus designed to measure waste output.

SUMMARY:
The purpose of this study is to test an electronic apparatus for measuring stool and urine output in an accurate and easy way. Participants will have one in-person or virtual visit with the study team prior to starting the study events. Participants that enroll in this study will have the freedom to choose when to begin and stop using the toilet apparatus when it is available for human testing. This apparatus will be located in a private bathroom in either the CIEMAS building or MSRB III Building.

ELIGIBILITY:
Inclusion Criteria:

* people who are able to use the private bathroom at no risk to themselves in the CIEMAS building (B508) or the bathroom located in room 4002, 4th floor of MSRB3.
* students or employees at Duke University since card access is required for our MSRB3 bathroom.
* people who spend most of their time in these buildings so we can assure the use of the toilet.
* If the recruitment number is slow, enrollment will include people from the closest buildings.

Exclusion Criteria:

* People who use wheelchairs or other mobility devices won't be able to enroll, since at this moment the bathroom is not compliant with the requirements on The Americans with Disabilities Act (ADA) of 1990.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of urine output correctly identified as measured by toilet seat apparatus . | Up to 3 months
  This analysis is intended to determine how accurately the apparatus measures urine output.
Percent of stool output correctly identified as measured by toilet seat apparatus . | Up to 3 months
  This analysis is intended to determine how accurately the apparatus measures stool output.

SECONDARY OUTCOMES:
Percent of urine weight correctly identified by toilet seat apparatus | Up to 3 months
  Measured by comparing participant weight loss before and after toilet use
Percent of stool weight correctly identified by toilet seat apparatus | Up to 3 months
  Measured by comparing participant weight loss before and after toilet use

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence David, Principal Investigator — Duke University - MGM
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No